CLINICAL TRIAL: NCT01856062
Title: Ovulation Induction With Clomiphene Citrate and Dexamethasone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeremy King, Reproductive Endocrinologist, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 379303-1
Record Dates: First submitted 2013-03-19; First posted 2013-05-17 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
Keywords: ovulation induction; dexamethasone
MeSH Terms: conditions — Infertility | interventions — Sugars; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene plus dexamethasone (Experimental): Oral dexamethasone will be added to clomiphene citrate
  Interventions: Drug: Dexamethasone
- Clomiphene plus placebo (Placebo Comparator): A placebo of dexamethasone will be given with clomiphene citrate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — A placebo with similar appearance to dexamethasone will be given with a standard regimen of clomiphene citrate (100mg/day oral for 5 days) for ovulation induction
  Other Names: sugar pill
  Arms: Clomiphene plus placebo
Drug: Dexamethasone — Oral dexamethasone will be added to a standard regimen of clomiphene citrate (100mg/day oral for 5 days) for ovulation induction
  Arms: Clomiphene plus dexamethasone

SUMMARY:
The purpose of this study is to determine if the addition of dexamethasone to clomiphene citrate will increase the pregnancy rate of intrauterine insemination (IUI) cycles.

DETAILED DESCRIPTION:
For decades clomiphene citrate (CC) has been the first line therapy for ovulation induction in anovulatory or oligoovulatory women, and for superovulation in women with unexplained infertility or partners with mild sperm abnormalities. While approximately 80% of patients achieve ovulation with CC, less than half conceive. Pregnancy is achieved in approximately 10% of ovulatory cycles.

Addition of dexamethasone to CC has been shown to result in pregnancy rates of 21-40% in CC-resistant women (defined as patients failing to ovulate on CC alone). A subsequent randomized controlled trial demonstrated higher pregnancy rates in patients with unexplained infertility undergoing intrauterine insemination (IUI) with CC + dexamethasone compared to those taking CC alone.

In light of the relatively high pregnancy rates achieved in previous trials, we hypothesize that dexamethasone as an adjunct to CC will increase the ovulation rate and pregnancy rate for all appropriate candidates for IU with a standard CC regimen.

Our study is designed to randomize patients undergoing ovulation induction with IUI into two groups: one consisting of a standard CC regimen, and the other consisting of the same CC regimen with the addition of daily dexamethasone. The primary outcome measure is pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military members or dependents seeking infertility treatment at Brooke Army Medical Center
* primary or secondary infertility
* candidate for intrauterine insemination (IUI)

Exclusion Criteria:

* Severe male factor infertility (total motile sperm count <10 million/mL)
* Bilateral fallopian tube obstruction
* Diminished ovarian reserve (baseline follicle stimulating hormone > 20)
* History of clomiphene resistance as determined by a Clomid challenge test or prior non-ovulatory cycles while taking clomiphene
* Known or suspected hypopituitarism or hypothalamic amenorrhea
* Six or more prior therapeutic CC cycles without a pregnancy
* Diabetes
* Renal impairment, hepatitis, hepatic cirrhosis, or myasthenia gravis
* Osteoporosis
* Cataracts or glaucoma
* Congenital Adrenal Hyperplasia, Cushing's disease, or any condition requiring chronic corticosteroid use

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 12 weeks
  Determined by serum hCG measurement

SECONDARY OUTCOMES:
Clinical pregnancy | 12 weeks
  Determined by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Massie, MD, Principal Investigator — San Antonio Military Medical Center
Locations (1):
- San Antonio Military Medical Center, Fort Sam Houston, Texas, United States